CLINICAL TRIAL: NCT03086330
Title: Efficacy and Safety of Semaglutide Once-weekly Versus Placebo as add-on to SGLT-2i in Subjects With Type 2 Diabetes Mellitus. A 30-week Randomised, Double-blind, Placebo-controlled Trial
Brief Title: Efficacy and Safety of Semaglutide Once-weekly Versus Placebo as add-on to SGLT-2i in Subjects With Type 2 Diabetes Mellitus
Acronym: SUSTAIN 9
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN9535-4269; 2016-000904-27 (EudraCT Number); U1111-1180-1213 (Other: WHO (World Health Organization)); JapicCTI-173542 (Registry Identifier: JAPIC)
Record Dates: First submitted 2017-03-14; First posted 2017-03-22 (Actual); Results first posted 2019-08-20 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-07

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Semaglutide (Experimental)
  Interventions: Drug: Semaglutide
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Semaglutide — Semaglutide, gradually increased to 1.0 mg, injected once weekly under the skin (subcutaneously, s.c.) for 30 weeks
  Arms: Semaglutide
Drug: Placebo — Semaglutide placebo, gradually increased to 1.0 mg, injected once weekly under the skin (subcutaneously, s.c.) for 30 weeks
  Arms: Placebo

SUMMARY:
This trial is conducted in Asia, Europe and North America. The aim of the trial is to compare the effect of semaglutide s.c. 1.0 mg once-weekly versus placebo as add-on to sodium glucose co-transporter-2 inhibitor (SGLT-2i) monotherapy or in combination with either metformin or sulfonylurea on glycaemic control after 30 weeks of treatment in subjects with type 2 diabetes. Subjects will remain on their pre-trial medication.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial
* Male or female, above or equal to 18 years at the time of signing informed consent. For Japan only: Male or female, age equal to or above 20 years at the time of signing informed consent
* Diagnosed with type 2 diabetes mellitus
* HbA1c of 7.0-10.0% (53-86 mmol/mol) (both inclusive)
* Stable dose of an SGLT-2 inhibitor as monotherapy or in combination (including fixed-dose drug combination) with a stable dose of metformin (equal to or above 1500 mg or maximum tolerated dose) or a SU for at least 90 days prior to the day of screening. All medications in compliance with current local label

Exclusion Criteria:

* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using an adequate contraceptive method (adequate contraceptive measure as required by local regulation or practice)
* Any disorder which in the investigator's opinion might jeopardise subject's safety or compliance with the protocol
* Treatment with any medication for the indication of diabetes or obesity other than stated in the inclusion criteria within the past 90 days prior to the day of screening. However, short term insulin treatment for a maximum of 14 days prior to the day of screening is allowed
* Subjects with alanine aminotransferase above 2.5 x upper normal limit
* Family or personal history of multiple endocrine neoplasia type 2 or medullary thyroid carcinoma. Family is defined as a first degree relative
* History or presence of pancreatitis (acute or chronic)
* History of diabetic ketoacidosis
* Any of the following: myocardial infarction, stroke, hospitalization for unstable angina or transient ischaemic attack within the past 180 days prior to the day of screening
* Subjects presently classified as being in New York Heart Association Class IV
* Planned coronary, carotid or peripheral artery revascularisation known on the day of screening
* Renal impairment measured as estimated Glomerular Filtration Rate value of eGFR below 60 ml/min/1.73 m^2 as defined by KDIGO 2012 classification using isotope dilution mass spectrometry for serum creatinine measured at screening
* Proliferative retinopathy or maculopathy requiring acute treatment. Verified by fundus photography or dilated fundoscopy performed within the past 90 days prior to randomisation
* Presence or history of malignant neoplasms within the past 5 years prior to the day of screening. Basal and squamous cell skin cancer and any carcinoma in-situ is allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2018-07-04 (Actual); Study Completion 2018-08-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (65):
- United States (41):
  - Novo Nordisk Investigational Site, Andalusia, Alabama
  - Novo Nordisk Investigational Site, Anniston, Alabama
  - Novo Nordisk Investigational Site, Glendale, Arizona
  - Novo Nordisk Investigational Site, Phoenix, Arizona
  - Novo Nordisk Investigational Site, Tempe, Arizona
  - Novo Nordisk Investigational Site, Little Rock, Arkansas
  - Novo Nordisk Investigational Site, La Jolla, California
  - Novo Nordisk Investigational Site, Lincoln, California
  - Novo Nordisk Investigational Site, Northridge, California
  - Novo Nordisk Investigational Site, Edgewater, Florida
  - Novo Nordisk Investigational Site, Maitland, Florida
  - Novo Nordisk Investigational Site, Lawrenceville, Georgia
  - Novo Nordisk Investigational Site, Woodstock, Georgia
  - Novo Nordisk Investigational Site, Hutchinson, Kansas
  - Novo Nordisk Investigational Site, Lexington, Kentucky
  - Novo Nordisk Investigational Site, Baltimore, Maryland
  - Novo Nordisk Investigational Site, Troy, Michigan
  - Novo Nordisk Investigational Site, Jefferson City, Missouri
  - Novo Nordisk Investigational Site, Albany, New York
  - Novo Nordisk Investigational Site, Smithtown, New York
  - Novo Nordisk Investigational Site, West Seneca, New York
  - Novo Nordisk Investigational Site, Charlotte, North Carolina
  - Novo Nordisk Investigational Site, Gastonia, North Carolina
  - Novo Nordisk Investigational Site, Greenville, North Carolina
  - Novo Nordisk Investigational Site, Kinston, North Carolina
  - Novo Nordisk Investigational Site, Morehead City, North Carolina
  - Novo Nordisk Investigational Site, Norman, Oklahoma
  - Novo Nordisk Investigational Site, Beaver, Pennsylvania
  - Novo Nordisk Investigational Site, McMurray, Pennsylvania
  - Novo Nordisk Investigational Site, Pittsburgh, Pennsylvania
  - Novo Nordisk Investigational Site, Arlington, Texas
  - Novo Nordisk Investigational Site, Austin, Texas
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Irving, Texas
  - Novo Nordisk Investigational Site, Shavano Park, Texas
  - Novo Nordisk Investigational Site, Sugar Land, Texas
  - Novo Nordisk Investigational Site, Victoria, Texas
  - Novo Nordisk Investigational Site, Murray, Utah
  - Novo Nordisk Investigational Site, Chesapeake, Virginia
  - Novo Nordisk Investigational Site, Olympia, Washington
- Austria (2):
  - Novo Nordisk Investigational Site, Saint Stefan
  - Novo Nordisk Investigational Site, Vienna
- Canada (7):
  - Novo Nordisk Investigational Site, Edmonton, Alberta
  - Novo Nordisk Investigational Site, Winnipeg, Manitoba
  - Novo Nordisk Investigational Site, Brampton, Ontario
  - Novo Nordisk Investigational Site, Etobicoke, Ontario
  - Novo Nordisk Investigational Site, Smiths Falls, Ontario
  - Novo Nordisk Investigational Site, Toronto, Ontario
  - Novo Nordisk Investigational Site, Waterloo, Ontario
- Japan (4):
  - Novo Nordisk Investigational Site, Kanagawa
  - Novo Nordisk Investigational Site, Nagakute-shi, Aichi
  - Novo Nordisk Investigational Site, Suita-shi, Osaka
  - Novo Nordisk Investigational Site, Tokyo
- Norway (7):
  - Novo Nordisk Investigational Site, Hamar
  - Novo Nordisk Investigational Site, Hoenefoss
  - Novo Nordisk Investigational Site, Namsos
  - Novo Nordisk Investigational Site, Olso
  - Novo Nordisk Investigational Site, Oslo
  - Novo Nordisk Investigational Site, Skedsmokorset
  - Novo Nordisk Investigational Site, Stavanger
- Novo Nordisk Investigational Site, Ponce, Puerto Rico
- Russia (3):
  - Novo Nordisk Investigational Site, Barnaul
  - Novo Nordisk Investigational Site, Novosibirsk
  - Novo Nordisk Investigational Site, Saint Petersburg

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com

REFERENCES:
- [Result] Zinman B, Bhosekar V, Busch R, Holst I, Ludvik B, Thielke D, Thrasher J, Woo V, Philis-Tsimikas A. Semaglutide once weekly as add-on to SGLT-2 inhibitor therapy in type 2 diabetes (SUSTAIN 9): a randomised, placebo-controlled trial. Lancet Diabetes Endocrinol. 2019 May;7(5):356-367. doi: 10.1016/S2213-8587(19)30066-X. Epub 2019 Mar 1. PMID 30833170

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 61 sites in 6 countries as follows: Austria (4 sites), Canada (8 sites), Japan (4 sites), Norway (4 sites), Russian Federation (5 sites), United States of America (USA) (36 sites). In addition, 1 site in Norway and 3 sites in the USA screened, but didn't randomise any participant.
Groups:
- Semaglutide 1.0 mg: Participants received semaglutide in a dose escalation manner for 30 weeks: 0.25 mg (weeks 1 to 4), 0.50 mg (weeks 5 to 8) and 1.0 mg (weeks 9 to 30). Semaglutide was taken once weekly as subcutaneous (s.c.) injections.
- Placebo: Participants received matching placebo (for semaglutide) in a dose escalation manner for 30 weeks. Placebo was taken once weekly as s.c. injections. Dose escalation for placebo matched that for semaglutide with regards to volume.
Period: Overall Study
Arm/Group | Semaglutide 1.0 mg | Placebo
Started | 151 | 151
Exposed | 150 | 151
Completed | 147 | 147
Not Completed | 4 | 4
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Semaglutide 1.0 mg: Participants received semaglutide in a dose escalation manner for 30 weeks: 0.25 mg (weeks 1 to 4), 0.50 mg (weeks 5 to 8) and 1.0 mg (weeks 9 to 30). Semaglutide was taken once weekly as s.c. injections.
- Total: Total of all reporting groups
Arm/Group | Semaglutide 1.0 mg | Placebo | Total
Number analyzed (Participants) | 151 | 151 | 302
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.5 (8.9) | 56.6 (10.1) | 57.0 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 64 | 126
  Male | 89 | 87 | 176
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 13 | 22
  Not Hispanic or Latino | 142 | 138 | 280
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska native | 2 | 0 | 2
  Asian | 36 | 35 | 71
  Black or African American | 9 | 4 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  White | 100 | 109 | 209
  Other | 4 | 3 | 7
Glycosylated haemoglobin (HbA1c) [Mean (Standard Deviation); unit: Percentage HbA1c] | 8.0 (0.8) | 8.1 (0.8) | 8.0 (0.8)

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c
Description: Change from baseline (week 0) in HbA1c was evaluated at week 30. Results are based on the 'on-treatment without rescue medication' observation period, which started at the date of first dose of trial product and ended at the first date of any of the following: 1) the last dose of trial product + 7 days or 2) initiation of rescue medication.
Time Frame: Week 0, week 30
Population: Full analysis set (FAS), which included all randomised participants. Number analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 151 | 151
Percentage of HbA1c | -1.6 (0.8) | -0.2 (0.9)
Statistical Analysis 1: Comparison: Semaglutide 1.0 mg vs Placebo; The responses were analysed using an analysis of covariance (ANCOVA) with treatment, stratification factor and region as fixed factors and baseline value as covariate. Before analysis, missing data were multiple imputed using observed data from participants within the same group defined by randomised treatment, using a regression model including stratification factor and region as categorical effects and data from baseline and all previous visits as covariates; Test type: Other; p < 0.0001, ANCOVA; Treatment difference = -1.42, 95% CI 2-sided [-1.61 to -1.24]

2. Secondary Outcome: Change in Body Weight (kg)
Description: Change from baseline (week 0) in body weight was evaluated at week 30. Results are based on the 'on-treatment without rescue medication' observation period.
Time Frame: Week 0, week 30
Population: FAS which included all randomised participants. Number analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 151 | 151
Kg | -4.7 (4.3) | -1.0 (3.1)
Statistical Analysis 1: Comparison: Semaglutide 1.0 mg vs Placebo; The responses were analysed using an ANCOVA with treatment, stratification factor and region as fixed factors and baseline value as covariate. Before analysis, missing data were multiple imputed using observed data from participants within the same group defined by randomised treatment, using a regression model including stratification factor and region as categorical effects and data from baseline and all previous visits as covariates; Test type: Other; p < 0.0001, ANCOVA; Treatment difference = -3.81, 95% CI 2-sided [-4.70 to -2.93]

3. Secondary Outcome: Change in Fasting Plasma Glucose (FPG)
Description: Change from baseline (week 0) in FPG was evaluated at week 30. Results are based on the 'on-treatment without rescue medication' observation period.
Time Frame: Week 0, week 30
Population: FAS which included all randomised participants. Number analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 151 | 151
mmol/L | -2.26 (2.05) | 0.07 (2.07)

4. Secondary Outcome: Change in Self-measured Plasma Glucose (SMPG), 7-point Profile: Mean 7-point Profile
Description: Change from baseline (week 0) in mean of the SMPG, 7-point profile was evaluated at week 30. Mean 7-point profile (the area under the profile) was calculated using the trapezoidal method and divided by the measurement time. Results are based on the 'on-treatment without rescue medication' observation period. Participants measured their plasma glucose at 7 different time points: before breakfast, 90 minutes after start of breakfast, before lunch, 90 minutes after start of lunch, before dinner, 90 minutes after start of dinner and at bedtime.
Time Frame: Week 0, week 30
Population: FAS which included all randomised participants. Number analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 151 | 151
mmol/L | -2.6 (1.9) | -0.3 (2.0)

5. Secondary Outcome: Change in Self-measured Plasma Glucose (SMPG), 7-point Profile: Mean Post Prandial Increment (Over All Meals)
Description: Change from baseline (week 0) in mean post prandial increment (over all meals) in the SMPG, 7-point profile was evaluated at week 30. The mean increment over all meals was derived as the mean of all available meal increments. Results are based on the 'on-treatment without rescue medication' observation period.
Time Frame: Week 0, week 30
Population: FAS which included all randomised participants. Number analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 151 | 151
mmol/L | -1.2 (2.0) | 0.0 (2.2)

6. Secondary Outcome: Change in Fasting Blood Lipid, Total Cholesterol
Description: Change from baseline (week 0) in total cholesterol (measured in mmol/L and presented as ratio to baseline) was evaluated at week 30. Results are based on the 'on-treatment without rescue medication' observation period.
Time Frame: Week 0, week 30
Population: FAS which included all randomised participants. Number analyzed = number of participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 151 | 151
Ratio | 0.91 (19.4) | 1.02 (18.9)

7. Secondary Outcome: Change in Fasting Blood Lipid, Low-density Lipoprotein (LDL) Cholesterol
Description: Change from baseline (week 0) in LDL (measured in mmol/L and presented as ratio to baseline) was evaluated at week 30. Results are based on the 'on-treatment without rescue medication' observation period.
Time Frame: Week 0, week 30
Population: FAS which included all randomised participants. Number analyzed = number of participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 151 | 151
Ratio | 0.90 (31.6) | 1.04 (27.7)

8. Secondary Outcome: Change in Fasting Blood Lipid, High-density Lipoprotein (HDL) Cholesterol
Description: Change from baseline (week 0) in HDL (measured in mmol/L and presented as ratio to baseline) was evaluated at week 30. Results are based on the 'on-treatment without rescue medication' observation period.
Time Frame: Week 0, week 30
Population: FAS which included all randomised participants. Number analyzed = number of participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 151 | 151
Ratio | 0.99 (15.8) | 1.01 (13.9)

9. Secondary Outcome: Change in Fasting Blood Lipid, Triglycerides
Description: Change from baseline (week 0) in triglycerides (measured in mmol/L and presented as ratio to baseline) was evaluated at week 30. Results are based on the 'on-treatment without rescue medication' observation period.
Time Frame: Week 0, week 30
Population: FAS which included all randomised participants. Number analyzed = number of participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 151 | 151
Ratio | 0.81 (41.3) | 0.97 (38.7)

10. Secondary Outcome: Change in Body Weight (%)
Description: Percent (%) change from baseline (week 0) in body weight (measured in kilogram (kg)) was evaluated at week 30. Results are based on the 'on-treatment without rescue medication' observation period.
Time Frame: Week 0, week 30
Population: FAS which included all randomised participants. Number analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 151 | 151
Percentage | -5.4 (4.8) | -1.0 (3.1)

11. Secondary Outcome: Change in Body Mass Index
Description: Change from baseline (week 0) in body mass index (BMI) was evaluated at week 30. Results are based on the 'on-treatment without rescue medication' observation period. BMI was calculated as 'body weight in kg/(height in meters) x (height in meters)'.
Time Frame: Week 0, week 30
Population: FAS which included all randomised participants. Number analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Kg/sqm
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 151 | 151
Kg/sqm | -1.7 (1.5) | -0.4 (1.1)

12. Secondary Outcome: Change in Waist Circumference
Description: Change from baseline (week 0) in waist circumference was evaluated at week 30. Results are based on the 'on-treatment without rescue medication' observation period.
Time Frame: Week 0, week 30
Population: FAS which included all randomised participants. Number analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 151 | 151
cm | -4.4 (5.5) | -1.8 (4.5)

13. Secondary Outcome: Change in Systolic Blood Pressure
Description: Change from baseline (week 0) in systolic blood pressure was evaluated at week 30. Results are based on the 'on-treatment without rescue medication' observation period.
Time Frame: Week 0, week 30
Population: FAS which included all randomised participants. Number analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 151 | 151
mmHg | -4.3 (14.5) | 1.1 (12.3)

14. Secondary Outcome: Change in Diastolic Blood Pressure
Description: Change from baseline (week 0) in diastolic blood pressure was evaluated at week 30. Results are based on the 'on-treatment without rescue medication' observation period.
Time Frame: Week 0, week 30
Population: FAS which included all randomised participants. Number analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 151 | 151
mmHg | -0.1 (8.1) | -0.1 (6.7)

15. Secondary Outcome: Change in Scores for Selected Patient Reported Outcomes: Short-form Health Survey (SF-36v2TM): Total Scores (Physical Component and Mental Component) and Scores From the 8 Domains
Description: Change from baseline (week 0) in patient reported outcome (PRO) questionnaire, SF-36v2TM was evaluated at week 30. The SF-36v2™ questionnaire was used to assess the overall health related quality of life of participants. This questionnaire contains 36 items and measures the individual overall health related quality of life on 8 domains: 1) Physical functioning, 2) Role functioning, 3) Bodily pain, 4) General health, 5) Vitality, 6) Social functioning, 7) Role emotional and 8) Mental health. Each item is scored on a scale from 1 to either 2, 3, 5, or 6; each item score is then converted to a scale of 0-100, representing the percentage of total possible score achieved and with higher scores indicating a higher health status; items on the same scale are then averaged to obtain the 8 scale scores. Physical component summary (PCS) includes domains 1-4 and mental component summary (MCS) includes domains 5-8. Higher PCS and MCS scores on a scale of 0-100 indicate a higher health status.
Time Frame: Week 0, week 30
Population: FAS which included all randomised participants. Number analyzed = number of participants with available data. Results are based on the 'on-treatment without rescue medication' observation period.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 151 | 151
Scores on a scale
  Physical component summary: number analyzed (Participants) | 117 | 125
  Physical component summary | 1.9 (4.9) | 0.7 (5.4)
  1) Physical functioning: number analyzed (Participants) | 117 | 125
  1) Physical functioning | 1.3 (4.1) | 1.1 (5.2)
  2) Role functioning: number analyzed (Participants) | 117 | 125
  2) Role functioning | 1.5 (6.1) | 0.0 (6.0)
  3) Bodily pain: number analyzed (Participants) | 117 | 125
  3) Bodily pain | 0.9 (7.4) | 0.1 (8.1)
  4) General health: number analyzed (Participants) | 117 | 125
  4) General health | 2.7 (6.8) | 0.1 (6.8)
  Mental component summary: number analyzed (Participants) | 117 | 125
  Mental component summary | 0.1 (5.6) | -0.9 (6.3)
  5) Vitality: number analyzed (Participants) | 117 | 125
  5) Vitality | 1.5 (6.2) | 0.2 (6.7)
  6) Social functioning: number analyzed (Participants) | 117 | 125
  6) Social functioning | 0.3 (7.3) | -1.0 (7.4)
  7) Role emotional: number analyzed (Participants) | 117 | 125
  7) Role emotional | 0.1 (6.7) | -0.2 (7.5)
  8) Mental health: number analyzed (Participants) | 117 | 125
  8) Mental health | 0.5 (5.2) | -0.6 (6.0)

16. Secondary Outcome: Change in Scores for Selected Patient Reported Outcomes: Diabetes Treatment Satisfaction Questionnaire (DTSQ): Treatment Satisfaction Score (Sum of 6 of 8 Items) and the 8 Items Separately
Description: Change from baseline (week 0) in PRO questionnaire, DTSQ was evaluated at week 30. Results are based on the 'on-treatment without rescue medication' observation period. The DTSQ measures satisfaction with diabetes treatment. The DTSQ consists of 8 items evaluating 6 aspects of treatment satisfaction and 2 perceived recent event rates of hyperglycemia/hypoglycemia. Each item is scored on a 7- point Likert scale ranging from 0 (very dissatisfied) to 6 (very satisfied). Items evaluating 6 aspects (items 3-8) of treatment satisfaction are summed to produce a total treatment satisfaction score; DTSQ status total scores range from 0-36, with higher scores indicating greater satisfaction; the perceived frequency of hyperglycemia/hypoglycemia items are scored separately, with lower scores indicating better perceived blood glucose control.
Time Frame: Week 0, week 30
Population: FAS which included all randomised participants. Number analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 151 | 151
Scores on a scale
  1) Feeling of unacceptably high blood sugars: number analyzed (Participants) | 119 | 125
  1) Feeling of unacceptably high blood sugars | -2.2 (1.9) | -0.8 (2.2)
  2) Feeling of unacceptably low blood sugars: number analyzed (Participants) | 119 | 125
  2) Feeling of unacceptably low blood sugars | 0.3 (1.5) | -0.4 (1.5)
  Total treatment satisfaction score (Sum of 3-8): number analyzed (Participants) | 119 | 125
  Total treatment satisfaction score (Sum of 3-8) | 4.2 (6.6) | 1.9 (7.0)
  3) Satisfaction with current treatment: number analyzed (Participants) | 119 | 125
  3) Satisfaction with current treatment | 0.8 (1.6) | 0.2 (1.4)
  4) Convenience of current treatment: number analyzed (Participants) | 119 | 125
  4) Convenience of current treatment | 0.7 (1.3) | 0.5 (1.3)
  5) Flexibility of current treatment: number analyzed (Participants) | 119 | 125
  5) Flexibility of current treatment | 0.7 (1.5) | 0.4 (1.7)
  6) Satisfaction with understanding of diabetes: number analyzed (Participants) | 119 | 125
  6) Satisfaction with understanding of diabetes | 0.5 (1.2) | 0.5 (1.5)
  7) Recommending treatment to others: number analyzed (Participants) | 119 | 125
  7) Recommending treatment to others | 0.8 (1.3) | 0.2 (1.8)
  8) Satisfaction to continue with present treatment: number analyzed (Participants) | 119 | 125
  8) Satisfaction to continue with present treatment | 0.8 (1.7) | 0.2 (1.7)

17. Secondary Outcome: HbA1c Below 7.0% (53 mmol/Mol)
Description: Percentage of participants with HbA1c below 7.0% (53 mmol/mol) was evaluated at week 30. Results are based on the 'on-treatment without rescue medication' observation period.
Time Frame: After 30 weeks
Population: FAS which included all randomised participants. Number analyzed = number of participants with available data.
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 120 | 127
Percentage of participants | 82.5 | 20.5

18. Secondary Outcome: HbA1c Equal to or Below 6.5% (48 mmol/Mol)
Description: Percentage of participants with HbA1c equal to or below 6.5% (48 mmol/mol) was evaluated at week 30. Results are based on the 'on-treatment without rescue medication' observation period.
Time Frame: After 30 weeks
Population: FAS which included all randomised participants. Number analyzed = number of participants with available data.
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 120 | 127
Percentage of participants | 60.0 | 3.9

19. Secondary Outcome: Weight Loss Equal to or Above 3%
Description: Percentage of participants with weight loss equal to or above 3% of their baseline (week 0) body weight was evaluated at week 30. Results are based on the 'on-treatment without rescue medication' observation period.
Time Frame: After 30 weeks
Population: FAS which included all randomised participants. Number analyzed = number of participants with available data.
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 121 | 128
Percentage of participants | 69.4 | 21.1

20. Secondary Outcome: Weight Loss Equal to or Above 5%
Description: Percentage of participants with weight loss equal to or above 5% of their baseline (week 0) body weight was evaluated at week 30. Results are based on the 'on-treatment without rescue medication' observation period.
Time Frame: After 30 weeks
Population: FAS which included all randomised participants. Number analyzed = number of participants with available data.
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 121 | 128
Percentage of participants | 50.4 | 7.8

21. Secondary Outcome: Weight Loss Equal to or Above 10%
Description: Percentage of participants with weight loss equal to or above 10% of their baseline (week 0) body weight was evaluated at week 30. Results are based on the 'on-treatment without rescue medication' observation period.
Time Frame: After 30 weeks
Population: FAS which included all randomised participants. Number analyzed = number of participants with available data.
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 121 | 128
Percentage of participants | 15.7 | 1.6

22. Secondary Outcome: HbA1c Below 7.0% (53 mmol/Mol) Without Severe or BG Confirmed Symptomatic Hypoglycaemia Episodes and no Weight Gain
Description: Percentage of participants with HbA1c below 7.0% (53 mmol/mol) without severe or BG confirmed symptomatic hypoglycaemia episodes and no weight gain from their baseline (week 0) body weight was evaluated at week 30. Severe or blood glucose (BG)-confirmed symptomatic hypoglycaemia: an episode that was severe according to the American Diabetes Association (ADA) classification or confirmed by a plasma glucose (PG) value below 3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia. Results are based on the 'on-treatment without rescue medication' observation period.
Time Frame: After 30 weeks
Population: FAS which included all randomised participants. Number analyzed = number of participants with available data.
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 120 | 127
Percentage of participants | 72.5 | 17.3

23. Secondary Outcome: HbA1c Reduction Equal to or Above 1%-Point
Description: Percentage of participants with HbA1c reduction equal to or above 1%-point was evaluated at week 30. Results are based on the 'on-treatment without rescue medication' observation period.
Time Frame: After 30 weeks
Population: FAS which included all randomised participants. Number analyzed = number of participants with available data.
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 120 | 127
Percentage of participants | 80.8 | 15.0

24. Secondary Outcome: HbA1c Reduction Equal to or Above 1%-Point and Weight Loss Equal to or Above 3%
Description: Percentage of participants with HbA1c reduction equal to or above 1%-point and weight loss equal to or above 3% of their baseline (week 0) body weight was evaluated at week 30. Results are based on the 'on-treatment without rescue medication' observation period.
Time Frame: After 30 weeks
Population: FAS which included all randomised participants. Number analyzed = number of participants with available data.
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 120 | 127
Percentage of participants | 56.7 | 7.9

25. Secondary Outcome: HbA1c Reduction Equal to or Above 1%-Point and Weight Loss Equal to or Above 5%
Description: Percentage of participants with HbA1c reduction equal to or above 1%-point and weight loss equal to or above 5% of their baseline (week 0) body weight was evaluated at week 30. Results are based on the 'on-treatment without rescue medication' observation period.
Time Frame: After 30 weeks
Population: FAS which included all randomised participants. Number analyzed = number of participants with available data.
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 120 | 127
Percentage of participants | 41.7 | 4.7

26. Secondary Outcome: HbA1c Reduction Equal to or Above 1%-Point and Weight Loss Equal to or Above 10%
Description: Percentage of participants with HbA1c reduction equal to or above 1%-point and weight loss equal to or above 10% of their baseline (week 0) body weight was evaluated at week 30. Results are based on the 'on-treatment without rescue medication' observation period.
Time Frame: After 30 weeks
Population: FAS which included all randomised participants. Number analyzed = number of participants with available data.
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 120 | 127
Percentage of participants | 15.0 | 1.6

27. Secondary Outcome: Number of Treatment-emergent Adverse Events (TEAEs)
Description: A TEAE was defined as an event that has onset date (or increase in severity) during the on-treatment observation period, which started at the date of first dose of trial product and ended at the last date on trial product + 42 days.
Time Frame: Week 0 - week 30
Population: Safety analysis set (SAS), which included all participants exposed to at least one dose of trial product (semaglutide or placebo).
Measure: Number; unit: Events
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 150 | 151
Events | 356 | 247

28. Secondary Outcome: Number of Treatment Emergent Severe or BG Confirmed Symptomatic Hypoglycaemic Episodes
Description: Hypoglycaemic episodes were defined as treatment emergent if the onset of the episode occurred within the on-treatment observation period, which started at the date of first dose of trial product and ended at the last date on trial product + 42 days. Severe or BG-confirmed symptomatic hypoglycaemia: an episode that was severe according to the ADA classification or confirmed by a PG value below 3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia.
Time Frame: Week 0 - week 30
Population: SAS, which included all participants exposed to at least one dose of trial product.
Measure: Number; unit: Episodes
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 150 | 151
Episodes | 4 | 0

29. Secondary Outcome: Change in Haematology: Haemoglobin
Description: Change from baseline (week 0) in haemoglobin was evaluated at week 30. Results are based on the on-treatment observation period, which started at the date of first dose of trial product and ended at the last date on trial product + 7 days.
Time Frame: Week 0, week 30
Population: SAS which included all participants exposed to at least one dose of trial product. Number analyzed = number of participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mmol/L
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 150 | 151
mmol/L | 1.1 (22.1) | 1.1 (29.3)

30. Secondary Outcome: Change in Haematology: Haematocrit
Description: Change from baseline (week 0) in haematocrit was evaluated at week 30. Results are based on the on-treatment observation period, which started at the date of first dose of trial product and ended at the last date on trial product + 7 days.
Time Frame: Week 0, week 30
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: % of red blood cells
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 150 | 151
% of red blood cells | 1.4 (130.3) | 1.1 (155.1)

31. Secondary Outcome: Change in Haematology: Thrombocytes
Description: Change from baseline (week 0) in thrombocytes was evaluated at week 30. Results are based on the on-treatment observation period, which started at the date of first dose of trial product and ended at the last date on trial product + 7 days.
Time Frame: Week 0, week 30
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 10^9 thrombocytes/L
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 150 | 151
10^9 thrombocytes/L | 25.3 (94.9) | 20.2 (100.7)

32. Secondary Outcome: Change in Haematology: Erythrocytes
Description: Change from baseline (week 0) in erythrocytes was evaluated at week 30. Results are based on the on-treatment observation period, which started at the date of first dose of trial product and ended at the last date on trial product + 7 days.
Time Frame: Week 0, week 30
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 10^12 erythrocytes/L
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 150 | 151
10^12 erythrocytes/L | 0.16 (111.0) | 0.11 (168.3)

33. Secondary Outcome: Change in Haematology: Leucocytes
Description: Change from baseline (week 0) in leucocytes was evaluated at week 30. Results are based on the on-treatment observation period, which started at the date of first dose of trial product and ended at the last date on trial product + 7 days.
Time Frame: Week 0, week 30
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 10^9 leucocytes/L
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 150 | 151
10^9 leucocytes/L | 0.65 (186.6) | 0.54 (146.8)

34. Secondary Outcome: Change in Biochemistry: Amylase
Description: Change from baseline (week 0) in amylase was evaluated at week 30. Results are based on the on-treatment observation period, which started at the date of first dose of trial product and ended at the last date on trial product + 7 days.
Time Frame: Week 0, week 30
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: U/L
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 150 | 151
U/L | 10.2 (113.8) | 5.0 (121.7)

35. Secondary Outcome: Change in Biochemistry: Lipase
Description: Change from baseline (week 0) in lipase was evaluated at week 30. Results are based on the on-treatment observation period, which started at the date of first dose of trial product and ended at the last date on trial product + 7 days.
Time Frame: Week 0, week 30
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: U/L
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 150 | 151
U/L | 11.6 (140.2) | 4.5 (171.8)

36. Secondary Outcome: Change in Biochemistry: Alkaline Phosphatase
Description: Change from baseline (week 0) in alkaline phosphatase was evaluated at week 30. Results are based on the on-treatment observation period, which started at the date of first dose of trial product and ended at the last date on trial product + 7 days.
Time Frame: Week 0, week 30
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: U/L
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 150 | 151
U/L | 4.6 (171.2) | 7.2 (106.7)

37. Secondary Outcome: Change in Biochemistry: Alanine Aminotransferase
Description: Change from baseline (week 0) in alanine aminotransferase was evaluated at week 30. Results are based on the on-treatment observation period, which started at the date of first dose of trial product and ended at the last date on trial product + 7 days.
Time Frame: Week 0, week 30
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: U/L
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 150 | 151
U/L | 4.5 (123.2) | 4.8 (166.7)

38. Secondary Outcome: Change in Biochemistry: Aspartate Aminotransferase
Description: Change from baseline (week 0) in aspartate aminotransferase was evaluated at week 30. Results are based on the on-treatment observation period, which started at the date of first dose of trial product and ended at the last date on trial product + 7 days.
Time Frame: Week 0, week 30
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: U/L
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 150 | 151
U/L | 3.4 (112.3) | 3.5 (90.1)

39. Secondary Outcome: Change in Biochemistry: Total Bilirubin
Description: Change from baseline (week 0) in total bilirubin was evaluated at week 30. Results are based on the on-treatment observation period, which started at the date of first dose of trial product and ended at the last date on trial product + 7 days.
Time Frame: Week 0, week 30
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: umol/L
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 150 | 151
umol/L | 2.3 (128.1) | 1.7 (134.8)

40. Secondary Outcome: Change in Biochemistry: Albumin
Description: Change from baseline (week 0) in albumin was evaluated at week 30. Results are based on the on-treatment observation period, which started at the date of first dose of trial product and ended at the last date on trial product + 7 days.
Time Frame: Week 0, week 30
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: g/dL
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 150 | 151
g/dL | 0.1 (45.4) | 0.1 (48.6)

41. Secondary Outcome: Change in Biochemistry: Calcium (Total)
Description: as for outcome 40
Time Frame: Week 0, week 30
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mmol/L
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 150 | 151
mmol/L | 0.04 (125.0) | 0.05 (88.9)

42. Secondary Outcome: Change in Biochemistry: Potassium
Description: Change from baseline (week 0) in potassium was evaluated at week 30. Results are based on the on-treatment observation period, which started at the date of first dose of trial product and ended at the last date on trial product + 7 days.
Time Frame: Week 0, week 30
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mmol/L
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 150 | 151
mmol/L | 0.3 (89.5) | 0.2 (73.7)

43. Secondary Outcome: Change in Biochemistry: Sodium
Description: Change from baseline (week 0) in sodium was evaluated at week 30. Results are based on the on-treatment observation period, which started at the date of first dose of trial product and ended at the last date on trial product + 7 days.
Time Frame: Week 0, week 30
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mmol/L
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 150 | 151
mmol/L | 1.7 (55.8) | 1.5 (48.4)

44. Secondary Outcome: Change in Biochemistry: Bicarbonate
Description: Change from baseline (week 0) in bicarbonate was evaluated at week 30. Results are based on the on-treatment observation period, which started at the date of first dose of trial product and ended at the last date on trial product + 7 days.
Time Frame: Week 0, week 30
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mmol/L
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 150 | 151
mmol/L | 2.2 (67.6) | 2.1 (69.0)

45. Secondary Outcome: Change in Biochemistry: Estimated Glomerular Filtration Rate (eGFR)
Description: Change from baseline (week 0) in eGFR was evaluated at week 30. Results are based on the on-treatment observation period, which started at the date of first dose of trial product and ended at the last date on trial product + 7 days.
Time Frame: Week 0, week 30
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min/1.73m2
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 150 | 151
mL/min/1.73m2 | 3.4 (114.8) | 3.2 (105.6)

46. Secondary Outcome: Change in Biochemistry: Creatinine
Description: Change from baseline (week 0) in creatinine was evaluated at week 30. Results are based on the on-treatment observation period, which started at the date of first dose of trial product and ended at the last date on trial product + 7 days.
Time Frame: Week 0, week 30
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: umol/L
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 150 | 151
umol/L | 4.6 (118.8) | 2.6 (191.5)

47. Secondary Outcome: Change in Calcitonin
Description: Change from baseline (week 0) in calcitonin was evaluated at week 30. Results are based on the on-treatment observation period, which started at the date of first dose of trial product and ended at the last date on trial product + 7 days.
Time Frame: Week 0, week 30
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/L
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 150 | 151
ng/L | 1.3 (172.1) | 1.7 (171.1)

48. Secondary Outcome: Change in Pulse
Description: Change from baseline (week 0) in pulse rate was evaluated at week 30. Results are based on the on-treatment observation period, which started at the date of first dose of trial product and ended at the last date on trial product + 7 days.
Time Frame: Week 0, week 30
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 150 | 151
beats/min | 4.0 (9.6) | 0.1 (8.4)

49. Secondary Outcome: Change in Electrocardiogram
Description: Electrocardiogram (ECG) results are presented for week 0 (baseline) and week 30. ECG finding are presented as percentage of participants with normal, abnormal non-clinically significant (NCS) and abnormal clinically significant (CS) ECG values. Results are based on the on-treatment observation period, which started at the date of first dose of trial product and ended at the last date on trial product + 42 days.
Time Frame: Week 0, week 30
Population: as for outcome 29
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 150 | 151
Percentage of participants
  Week 0: Normal: number analyzed (Participants) | 149 | 151
  Week 0: Normal | 62.4 | 66.2
  Week 0: Abnormal, NCS: number analyzed (Participants) | 149 | 151
  Week 0: Abnormal, NCS | 36.9 | 32.5
  Week 0: Abnormal, CS: number analyzed (Participants) | 149 | 151
  Week 0: Abnormal, CS | 0.7 | 1.3
  Week 30: Normal: number analyzed (Participants) | 129 | 143
  Week 30: Normal | 64.3 | 66.4
  Week 30: Abnormal, NCS: number analyzed (Participants) | 129 | 143
  Week 30: Abnormal, NCS | 34.9 | 32.2
  Week 30: Abnormal, CS: number analyzed (Participants) | 129 | 143
  Week 30: Abnormal, CS | 0.8 | 1.4

50. Secondary Outcome: Change in Physical Examination: General Appearance
Description: Physical examination (general appearance) results are presented for week -2 (baseline) and week 30. Results are presented as percentage of participants with normal, abnormal NCS and abnormal CS findings. Results are based on the on-treatment observation period, which started at the date of first dose of trial product and ended at the last date on trial product + 7 days.
Time Frame: Week -2, week 30
Population: as for outcome 29
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 150 | 151
Percentage of participants
  Week -2: Normal: number analyzed (Participants) | 150 | 150
  Week -2: Normal | 90.0 | 86.0
  Week -2: Abnormal, NCS: number analyzed (Participants) | 150 | 150
  Week -2: Abnormal, NCS | 10.0 | 14.0
  Week -2: Abnormal, CS: number analyzed (Participants) | 150 | 150
  Week -2: Abnormal, CS | 0 | 0
  Week 30: Normal: number analyzed (Participants) | 121 | 139
  Week 30: Normal | 87.6 | 87.1
  Week 30: Abnormal, NCS: number analyzed (Participants) | 121 | 139
  Week 30: Abnormal, NCS | 11.6 | 12.2
  Week 30: Abnormal, CS: number analyzed (Participants) | 121 | 139
  Week 30: Abnormal, CS | 0.8 | 0.7

51. Secondary Outcome: Change in Physical Examination: Central and Peripheral Nervous System
Description: Physical examination (central and peripheral nervous system) results are presented for week -2 (baseline) and week 30. Results are presented as percentage of participants with normal, abnormal NCS and abnormal CS findings. Results are based on the on-treatment observation period, which started at the date of first dose of trial product and ended at the last date on trial product + 7 days.
Time Frame: Week -2, week 30
Population: as for outcome 29
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 150 | 151
Percentage of participants
  Week -2: Normal: number analyzed (Participants) | 150 | 150
  Week -2: Normal | 92.0 | 86.7
  Week -2: Abnormal, NCS: number analyzed (Participants) | 150 | 150
  Week -2: Abnormal, NCS | 7.3 | 12.7
  Week -2: Abnormal, CS: number analyzed (Participants) | 150 | 150
  Week -2: Abnormal, CS | 0.7 | 0.7
  Week 30: Normal: number analyzed (Participants) | 121 | 139
  Week 30: Normal | 94.2 | 87.8
  Week 30: Abnormal, NCS: number analyzed (Participants) | 121 | 139
  Week 30: Abnormal, NCS | 5.0 | 12.2
  Week 30: Abnormal, CS: number analyzed (Participants) | 121 | 139
  Week 30: Abnormal, CS | 0.8 | 0

52. Secondary Outcome: Change in Physical Examination: Cardiovascular System
Description: Physical examination (cardiovascular system) results are presented for week -2 (baseline) and week 30. Results are presented as percentage of participants with normal, abnormal NCS and abnormal CS findings. Results are based on the on-treatment observation period, which started at the date of first dose of trial product and ended at the last date on trial product + 7 days.
Time Frame: Week -2, week 30
Population: as for outcome 29
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 150 | 151
Percentage of participants
  Week -2: Normal: number analyzed (Participants) | 150 | 150
  Week -2: Normal | 98.7 | 93.3
  Week -2: Abnormal, NCS: number analyzed (Participants) | 150 | 150
  Week -2: Abnormal, NCS | 1.3 | 6.0
  Week -2: Abnormal, CS: number analyzed (Participants) | 150 | 150
  Week -2: Abnormal, CS | 0 | 0.7
  Week 30: Normal: number analyzed (Participants) | 121 | 139
  Week 30: Normal | 98.3 | 92.8
  Week 30: Abnormal, NCS: number analyzed (Participants) | 121 | 139
  Week 30: Abnormal, NCS | 1.7 | 7.2
  Week 30: Abnormal, CS: number analyzed (Participants) | 121 | 139
  Week 30: Abnormal, CS | 0 | 0

53. Secondary Outcome: Change in Physical Examination: Gastrointestinal System Including Mouth
Description: Physical examination (gastrointestinal system including mouth) results are presented for week -2 (baseline) and week 30. Results are presented as percentage of participants with normal, abnormal NCS and abnormal CS findings. Results are based on the on-treatment observation period, which started at the date of first dose of trial product and ended at the last date on trial product + 7 days.
Time Frame: Week -2, week 30
Population: as for outcome 29
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 150 | 151
Percentage of participants
  Week -2: Normal: number analyzed (Participants) | 150 | 150
  Week -2: Normal | 93.3 | 93.3
  Week -2: Abnormal, NCS: number analyzed (Participants) | 150 | 150
  Week -2: Abnormal, NCS | 6.7 | 6.7
  Week -2: Abnormal, CS: number analyzed (Participants) | 150 | 150
  Week -2: Abnormal, CS | 0 | 0
  Week 30: Normal: number analyzed (Participants) | 121 | 139
  Week 30: Normal | 95.9 | 94.2
  Week 30: Abnormal, NCS: number analyzed (Participants) | 121 | 139
  Week 30: Abnormal, NCS | 3.3 | 5.8
  Week 30: Abnormal, CS: number analyzed (Participants) | 121 | 139
  Week 30: Abnormal, CS | 0.8 | 0

54. Secondary Outcome: Change in Physical Examination: Skin
Description: Physical examination (skin) results are presented for week -2 (baseline) and week 30. Results are presented as percentage of participants with normal, abnormal NCS and abnormal CS findings. Results are based on the on-treatment observation period, which started at the date of first dose of trial product and ended at the last date on trial product + 7 days.
Time Frame: Week -2, week 30
Population: as for outcome 29
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 150 | 151
Percentage of participants
  Week -2: Normal: number analyzed (Participants) | 150 | 150
  Week -2: Normal | 91.3 | 93.3
  Week -2: Abnormal, NCS: number analyzed (Participants) | 150 | 150
  Week -2: Abnormal, NCS | 8.7 | 6.7
  Week -2: Abnormal, CS: number analyzed (Participants) | 150 | 150
  Week -2: Abnormal, CS | 0 | 0
  Week 30: Normal: number analyzed (Participants) | 121 | 139
  Week 30: Normal | 93.4 | 95.0
  Week 30: Abnormal, NCS: number analyzed (Participants) | 121 | 139
  Week 30: Abnormal, NCS | 6.6 | 4.3
  Week 30: Abnormal, CS: number analyzed (Participants) | 121 | 139
  Week 30: Abnormal, CS | 0 | 0.7

55. Secondary Outcome: Change in Physical Examination: Respiratory System
Description: Physical examination (respiratory system) results are presented for week -2 (baseline) and week 30. Results are presented as percentage of participants with normal, abnormal NCS and abnormal CS findings. Results are based on the on-treatment observation period, which started at the date of first dose of trial product and ended at the last date on trial product + 7 days.
Time Frame: Week -2, week 30
Population: as for outcome 29
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 150 | 151
Percentage of participants
  Week -2: Normal: number analyzed (Participants) | 150 | 150
  Week -2: Normal | 100 | 98.7
  Week -2: Abnormal, NCS: number analyzed (Participants) | 150 | 150
  Week -2: Abnormal, NCS | 0 | 1.3
  Week -2: Abnormal, CS: number analyzed (Participants) | 150 | 150
  Week -2: Abnormal, CS | 0 | 0
  Week 30: Normal: number analyzed (Participants) | 121 | 139
  Week 30: Normal | 100 | 99.3
  Week 30: Abnormal, NCS: number analyzed (Participants) | 121 | 139
  Week 30: Abnormal, NCS | 0 | 0.7
  Week 30: Abnormal, CS: number analyzed (Participants) | 121 | 139
  Week 30: Abnormal, CS | 0 | 0

56. Secondary Outcome: Change in Physical Examination: Lymph Node Palpation
Description: Physical examination (lymph node palpation) results are presented for week -2 (baseline) and week 30. Results are presented as percentage of participants with normal, abnormal NCS and abnormal CS findings. Results are based on the on-treatment observation period, which started at the date of first dose of trial product and ended at the last date on trial product + 7 days.
Time Frame: Week -2, week 30
Population: as for outcome 29
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 150 | 151
Percentage of participants
  Week -2: Normal: number analyzed (Participants) | 150 | 150
  Week -2: Normal | 99.3 | 100
  Week -2: Abnormal, NCS: number analyzed (Participants) | 150 | 150
  Week -2: Abnormal, NCS | 0.7 | 0
  Week -2: Abnormal, CS: number analyzed (Participants) | 150 | 150
  Week -2: Abnormal, CS | 0 | 0
  Week 30: Normal: number analyzed (Participants) | 121 | 139
  Week 30: Normal | 99.2 | 100
  Week 30: Abnormal, NCS: number analyzed (Participants) | 121 | 139
  Week 30: Abnormal, NCS | 0 | 0
  Week 30: Abnormal, CS: number analyzed (Participants) | 121 | 139
  Week 30: Abnormal, CS | 0.8 | 0

57. Secondary Outcome: Change in Physical Examination: Thyroid Gland
Description: Physical examination (thyroid gland) results are presented for week -2 (baseline) and week 30. Results are presented as percentage of participants with normal, abnormal NCS and abnormal CS findings. Results are based on the on-treatment observation period, which started at the date of first dose of trial product and ended at the last date on trial product + 7 days.
Time Frame: Week -2, week 30
Population: as for outcome 29
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 150 | 151
Percentage of participants
  Week -2: Normal: number analyzed (Participants) | 150 | 150
  Week -2: Normal | 98.0 | 96.7
  Week -2: Abnormal, NCS: number analyzed (Participants) | 150 | 150
  Week -2: Abnormal, NCS | 2.0 | 3.3
  Week -2: Abnormal, CS: number analyzed (Participants) | 150 | 150
  Week -2: Abnormal, CS | 0 | 0
  Week 30: Normal: number analyzed (Participants) | 121 | 139
  Week 30: Normal | 99.2 | 97.1
  Week 30: Abnormal, NCS: number analyzed (Participants) | 121 | 139
  Week 30: Abnormal, NCS | 0.8 | 2.9
  Week 30: Abnormal, CS: number analyzed (Participants) | 121 | 139
  Week 30: Abnormal, CS | 0 | 0

58. Secondary Outcome: Change in Fundoscopy
Description: Fundoscopy results for both left and right eyes are presented for week 0 (baseline) and week 30. Results are presented as percentage of participants with normal, abnormal NCS and abnormal CS findings. Results are based on the on-treatment observation period, which started at the date of first dose of trial product and ended at the last date on trial product + 7 days.
Time Frame: Week 0, week 30
Population: as for outcome 29
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 150 | 151
Percentage of participants
  Left eye: Week 0; normal: number analyzed (Participants) | 150 | 150
  Left eye: Week 0; normal | 70.7 | 62.0
  Left eye: Week 0; abnormal, NCS: number analyzed (Participants) | 150 | 150
  Left eye: Week 0; abnormal, NCS | 24.7 | 32.7
  Left eye: Week 0; abnormal, CS: number analyzed (Participants) | 150 | 150
  Left eye: Week 0; abnormal, CS | 4.7 | 5.3
  Left eye: Week 30; normal: number analyzed (Participants) | 82 | 92
  Left eye: Week 30; normal | 79.3 | 64.1
  Left eye: Week 30; abnormal, NCS: number analyzed (Participants) | 82 | 92
  Left eye: Week 30; abnormal, NCS | 17.1 | 31.5
  Left eye: Week 30; abnormal, CS: number analyzed (Participants) | 82 | 92
  Left eye: Week 30; abnormal, CS | 3.7 | 4.3
  Right eye: Week 0; normal: number analyzed (Participants) | 150 | 149
  Right eye: Week 0; normal | 69.3 | 62.4
  Right eye: Week 0; abnormal, NCS: number analyzed (Participants) | 150 | 149
  Right eye: Week 0; abnormal, NCS | 25.3 | 30.9
  Right eye: Week 0; abnormal, CS: number analyzed (Participants) | 150 | 149
  Right eye: Week 0; abnormal, CS | 5.3 | 6.7
  Right eye: Week 30; normal: number analyzed (Participants) | 82 | 91
  Right eye: Week 30; normal | 75.6 | 63.7
  Right eye: Week 30; abnormal, NCS: number analyzed (Participants) | 82 | 91
  Right eye: Week 30; abnormal, NCS | 19.5 | 31.9
  Right eye: Week 30; abnormal, CS: number analyzed (Participants) | 82 | 91
  Right eye: Week 30; abnormal, CS | 4.9 | 4.4

ADVERSE EVENTS:
Time Frame: Week 0 to week 30 (treatment period) + 42 days (follow-up period). All the reported adverse events (AEs) are TEAEs.
Description: Results are based on the SAS. Treatment with semaglutide or placebo followed a fixed dose escalation. The maintenance dose of semaglutide 1.0 mg was reached after 4 doses (4 weeks) of 0.25 mg, followed by 4 doses (4 weeks) of 0.5 mg. The same fixed dose escalation scheme was followed for placebo, with respective dose matching volume. Hence, the adverse events are combinedly presented under 2 respective reporting groups, 'semaglutide 1.0 mg and placebo'.
Arm/Group | Semaglutide 1.0 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/150 | 0/151
Serious Adverse Events (participants affected / at risk) | 7/150 | 6/151
Other Adverse Events (participants affected / at risk) | 49/150 | 28/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide 1.0 mg (N=150) | Placebo (N=151)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Gastroenteritis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Neurocysticercosis (Infections and infestations) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Retinal artery occlusion (Eye disorders) | 1 (1) | 0 (0)
Thyroidectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide 1.0 mg (N=150) | Placebo (N=151)
Constipation (Gastrointestinal disorders) | 10 (10) | 0 (0)
Diabetic retinopathy (Eye disorders) | 2 (2) | 8 (9)
Diarrhoea (Gastrointestinal disorders) | 17 (21) | 9 (11)
Nasopharyngitis (Infections and infestations) | 8 (9) | 8 (11)
Nausea (Gastrointestinal disorders) | 29 (37) | 5 (7)
Vomiting (Gastrointestinal disorders) | 14 (21) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-18): https://cdn.clinicaltrials.gov/large-docs/30/NCT03086330/Prot_SAP_000.pdf